CLINICAL TRIAL: NCT05010551
Title: Translation and Validation of Modified Polycystic Ovary Syndrome Questionnaire in Urdu Language
Brief Title: Translation and Validation of MPCOSQ in Urdu Language
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00843 Rabbiya Zaman
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: PCOS- Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To translate and validate modifies polycystic ovary syndrome quality of life (MPCOQ) questionnaire into Urdu. To evaluate the reliability, validity and of Urdu version of modified polycystic ovary syndrome quality of life questionnaire (MPCOQ).

DETAILED DESCRIPTION:
* All statistical analyses will be conducted using the Statistical Product and Service Solution version 21 software.
* Continuous variables will be shown by mean and standard deviation and the categories will be demonstrated in frequency and percentage.
* In this study, factor structure of the (MPCOQ) will be analyzed using the principal component factor analysis with varimax rotation.
* Intraclass Correlation Coefficient (ICC) (95% confidence interval) will be used for test-retest value and Cronbach's Alpha will be used for internal consistency analysis.
* Measurement error will be determined by calculating the standard error of measurement (SEM) and the Smallest Detectable Change (SDC). Independent t-test will be used to determine the differences between groups

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 - 30

  * Married
  * Female patients diagnosed with PCOS, having 2 of the following Rotterdam diagnostic criteria:

I. Polycystic ovaries visualized on ultrasound scan (presence of 12 follicles or more in one or both ovaries and/or increased ovarian volume >10ml II. Clinical signs of hyperandrogenism (the hirsutism score based on the Ferriman-Gallwey score >7 or obvious acne) III. Having an interval between menstrual periods >35 days and/or amenorrhea as the absence of vaginal bleeding for at least 6 months, i.e. 199 days Patients who are willing to participate

Exclusion Criteria:

* • Non-adrenal hyperplasia, thyroid dysfunction, and hyperprolactinemia

  * Female undergoing Hormone Replacement Therapy
  * Female with malignancies
  * Any recent fractures, surgeries
  * Patient with nephrological and neurological conditions
  * Dementia or cognitive impairments

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Married Diagnosed with PCOS
Study Population: Patients diagnosed with PCOS
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Modified polycystic ovary syndrome quality of life questionnaire | 6 months
  The tool is to measure health related quality of life of females suffering from PCOS. it contains 30 items with 6 main areas related to hirsutism , acne, weight, infertility, emotional disturbance, menstrual difficulties to define different symptoms of PCOS. then quality of life will be measured of respective patients. The total is 210 with higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, Principal Investigator — Riphah International University; Abeer Fatima, MS(cppt), Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Abeer Fatima, Islamabad, Punjab Province
  - Zohra Institute of Health Sciences, Rawalpindi

IPD SHARING:
Plan to Share IPD: No